CLINICAL TRIAL: NCT03122951
Title: Clearblue® Advanced Ovulation Test User Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROTOCOL-0917
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-09

CONDITIONS: Trying to Conceive Population

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ovulation test use (Other): All voluteers will receive device for use according to instructions
  Interventions: Diagnostic Test: ovulation test use

INTERVENTIONS:
Diagnostic Test: ovulation test use — Normal use of The Clearblue® Advanced Ovulation Test according to Information for use instructions

SUMMARY:
The Clearblue® Advanced Ovulation Test is designed for home use by women who are either planning or trying for a pregnancy.

The purpose of this protocol is to demonstrate that lay-users representative of the target user population are able to use the product in the intended user environment.

DETAILED DESCRIPTION:
The Clearblue Advanced Ovulation Test is designed for home use by women who are trying to get pregnant now or in the near future. It identifies those days in a woman's cycle on which intercourse is most likely to lead to conception.

The product defines three phases of fertility through urine hormone measurement: Low (small chance of conceiving), High (increased chance of conceiving) which is achieved by the detection of a rise in the level of estrone-3-glucuronide and Peak (highest chance of conceiving) which provides an early warning of impending ovulation through detection of the luteinising hormone surge which precedes it by 24 - 36 hours.

This protocol aims to demonstrate the successful usage of the Clearblue Advanced Ovulation Test product by lay-users in the intended environment.

Elements of system usability, product satisfaction and ease of use will be used to assess overall product performance in lay-user hands.

Lay users will be required to user the product according to the instructions for use for a mimimum of 1 complete menstrual cycle after which they will be required to provide feedback on product use.

A usability scale which focusses on providing subjective feedback from users. This is a simple ten-item attitude Likert scale which each volunteer will complete after 4 weeks of product use. The primary endpoints of this study will focus on the use of this scoring scale to determine the usability of the product in lay-user hands.

ELIGIBILITY:
Inclusion Criteria:

Female Aged 18 to 45 years Trying to conceive, planning to conceive in the next year or interested in using an ovulation testing system.

Willing to provide written informed consent to participate in the study. Has menstrual cycles.

Exclusion Criteria:

Pregnant, recently pregnant or breastfeeding Diagnosed with Polycystic Ovarian Syndrome Use of hormonal contraception Use of hormone replacement therapy Use of any other medical treatment for fertility such as ovulation drugs, artificial insemination, assisted fertility such as IVF, ICSI Currently or previously employed by SPD, Alere, Unipath or P and G, or affiliates Has an immediate relative currently or previously employed by SPD, Alere, Unipath or P and G or affiliates

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 577 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
proportion of users who score the product above average according to the system usability score after 4 weeks of usage | 4 weeks
  ≥95% of volunteers score 68 or higher on the usability scale after 4 weeks of usage or at the point of withdrawal from the study

SECONDARY OUTCOMES:
agreement between lay-user interpretation of the test result and the test result as stored in the users account | 4 weeks
  agreement between lay-user interpretation of the test result and the test result as stored in the users account
Within and between volunteer experience of using the product | 4 weeks
  Intra and inter-volunteer experience of using the product as recorded on a satisfaction scale in the volunteer diary
level of lay-user interaction with the product | 4 weeks
  The average number of times an individual volunteer interacts with the product throughout a cycle and an understanding of when the interaction is at its highest
Product ease of use and comprehension of instructions for use | 4 weeks
  The cumulative Likert scored for the end of study system usability questions

CONTACTS AND LOCATIONS:
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No